CLINICAL TRIAL: NCT07152184
Title: A Prospective, Randomized, and Controlled Study Comparing Two Treatment Strategies (Dose REduction of Antipsychotics vs. Maintenance Treatment) in Patients With Schizophrenia Spectrum Disorder After Stratification Based on Patients' Psychotic PHENotype: a Personalized Medicine Approach
Brief Title: Study Comparing Antipsychotic Dose Reduction vs. Maintenance Treatment in Patients With Schizophrenia Spectrum Disorder: a Personalized Medicine Approach
Acronym: DREAMS-Phen
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8669; 2023-509558-80-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Patient With Schizophrenia Spectrum Disorder; NLM Classification WM 203, Psychology:Schizophrenic Psychology; Schizophrenia Spectrum and Other Psychotic Disorders
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients with Cycloid Psychosis receiving the Dose Reduction strategy (CP-DR) (Experimental): After verifying the patient's phenotype, only those with cycloid psychosis will be included in this arm. The patient's usual antipsychotic dose will be gradually reduced to doses lower than those recommended by the marketing authorization (AMM).
  Interventions: Drug: Use of antipsychotic treatment with marketing authorization at doses lower than those recommended: - Olanzapine - Zuclopenthixol - Risperidone - Pipotiazine palmitate / Pipotiazine - Quetiapine - Flup
- Patients with Cycloid Psychosis receiving the Maintenance Treatment strategy (CP-MT) (Active Comparator): After verifying the patient's phenotype, only those with cycloid psychosis will be included in this arm. The patient's usual antipsychotic dose will be maintained in accordance with those recommended by the marketing authorization (AMM).
  Interventions: Drug: Use of antipsychotic treatment with marketing authorization at doses lower than those recommended: - Olanzapine - Zuclopenthixol - Risperidone - Pipotiazine palmitate / Pipotiazine - Quetiapine - Flup
- Patients with Non-Cycloid Psychosis receiving the Dose Reduction strategy (Non-CP-DR) (Experimental): After verifying the patient's phenotype, only those without cycloid psychosis will be included in this arm. The patient's usual antipsychotic dose will be gradually reduced to doses lower than those recommended by the marketing authorization (AMM).
  Interventions: Drug: Use of antipsychotic treatment with marketing authorization at doses lower than those recommended: - Olanzapine - Zuclopenthixol - Risperidone - Pipotiazine palmitate / Pipotiazine - Quetiapine - Flup
- patients with Non-Cycloid Psychosis receiving the Maintenance Treatment strategy (Non-CP-MT) (Active Comparator): After verifying the patient's phenotype, only those without cycloid psychosis will be included in this arm. The patient's usual antipsychotic dose will be maintained in accordance with those recommended by the marketing authorization (AMM).
  Interventions: Drug: Use of antipsychotic treatment with marketing authorization at doses lower than those recommended: - Olanzapine - Zuclopenthixol - Risperidone - Pipotiazine palmitate / Pipotiazine - Quetiapine - Flup

INTERVENTIONS:
Drug: Use of antipsychotic treatment with marketing authorization at doses lower than those recommended: - Olanzapine - Zuclopenthixol - Risperidone - Pipotiazine palmitate / Pipotiazine - Quetiapine - Flup — Biological A blood sample of up to 5 mL will be taken at visits V0, V5, and V14, for a maximum total volume of 15 mL for the study.
  Behavioral Quality of life and disease assessment questionnaires will need to be completed by the patient and their caregiver.

SUMMARY:
The objective of this study is to respond to frequent requests from patients who wish to reduce or even stop their antipsychotic treatment once they have achieved clinical stability. Psychiatrists are reluctant to respond to these requests because the method for safely reducing or stopping antipsychotic treatment remains poorly understood.

The investigators want to verify the existence of an interaction between treatment strategy and psychotic phenotype (cycloid psychosis vs. non-CP), i.e., in terms of functional remission, the benefit of the dose reduction strategy compared to the maintenance strategy will be greater in the CP group than in the non-CP group.

To this end, patients will be randomly assigned to four groups based on their phenotype and treatment strategy (CP-dose reduction; CP-dose maintenance; non-CP-dose reduction; and non-CP-dose maintenance).

Several hospitals throughout France are participating in this study, in which a random draw (called randomization) will be conducted to determine whether the physician will propose reducing the antipsychotic dose or maintaining it at the same dose for the patient.

Patients included in this study will be adults aged 18 to 60 who have been diagnosed with a schizophrenic spectrum disorder (SS): schizophrenia, schizophreniform disorder, schizoaffective disorder, or brief psychotic episode.

The antipsychotics studied are:

* second-generation antipsychotics: amisulpride, aripiprazole, olanzapine, quetiapine, risperidone;
* first-generation antipsychotics: chlorpromazine, flupentixol, haloperidol, levomepromazine, loxapine, pipotiazine, zuclopenthixol.

  288 patients will be included and followed for 24 months. The inclusion period is 48 months.

Fourteen follow-up visits are planned, every month for four months and then every two months. During these visits, self-questionnaires or cognitive tests will have to be completed by the patient, the caregiver, and/or the treating psychiatrist.

Three blood samples will be taken at inclusion, at 6 months, and at the end of the study, in particular to measure the level of medication in the blood.

ELIGIBILITY:
Inclusion Criteria:

* - Patient 18-60 years of age;
* Patient affiliated to health insurance (beneficiary or beneficiary's family);
* Patient informed of the results of the preliminary medical examination;
* Patient able to understand the aims and risks of the research (assisted by his/her curator, if applicable (if subject under curatorship*))
* Informed consent signed by patient
* Patient with a diagnosis of schizophrenia spectrum disorder (SSD): schizophrenia, schizophreniform, schizoaffective disorder or brief psychotic episode according to DSM-5;
* Patient with:

  1. Either a cycloid psychosis (CP) phenotype according to By-CP (score >=80%)
  2. Or another (non-CP) psychotic phenotype; (By-CP score < 80%)
* Outpatient followed by an ambulatory psychiatrist;
* Patient with an identified caregiver, defined as a person able to support the patient for the duration of the study, spending at least 8 hours per week with the patient or having easy access to the patient per phone.
* Patient clinically stabilized, for at least 6 months, as defined by

  a) low intensity of positive symptoms, i.e. PANSS P1, P2 and P3 items < 4.
* Patient treated with oral antipsychotics (in mono or polytherapy, with second- or first-generation antipsychotics);
* Patients with a PSP score >70 at baseline will also be included
* The participant agrees to follow the contraceptive requirements detailed in the protocol *Subjects under limited guardianship (i.e. French "curatelle") can participate to the study.

Exclusion Criteria:

* - Patient hospitalized in a psychiatric ward;
* Patient with a recent psychotic episode (during the last 6 months);
* Patient treated with long-acting injection of antipsychotics (due to feasibility constraints and to the fact that these treatments remain essentially proposed to non-compliant patients with high risk of acute cessation and loss to follow-up);
* Patient treated with clozapine (in mono or polytherapy - highly resistant patients, specificities of the relapses under clozapine
* Patient considered by his psychiatrists to be at serious risk of harm to self or others (e.g. previous aggressive or suicidal behaviors); notably, a patient answering "yes" to C-SSRS suicidal ideation Type 4 or 5, having any suicidal behavior assessment within 6 months at Screening, or having been hospitalized or treated for suicidal behavior in the past 5 years before Screening. The investigator will rely on the results of the C-SSRS questionnaire completed at the time of inclusion (after consent has been signed) or previously completed as part of the patient's follow-up according to current practice.
* Neurological or severe medical condition other than psychosis;
* Pregnancy (verified by urinary test at enrollment for women of childbearing potential);
* Current breastfeeding;
* Patient involved in another Investigational Medicinal Product trial or having participated in another investigational drug trial, in which they received the investigational drug, within 60 days
* Patient in an exclusion period defined by another research protocol;
* Patient under guardianship (i.e. French 'tutelle');
* Patient with care under constraint
* Patients deprived of freedom because of a judicial measure.
* Inability to give the patient the written consent form (emergency situation)
* Patients with major depressive disorder (CDSS > 5) or manic episode (DSM-5-TR)
* Patients with any of the following signs of substance abuse:

  1. Current diagnosis or history of substance use disorder and/or substance intoxication as defined in the DSM-5-TR. If the history of substance use disorder is more than 12 months before baseline, the participant may be allowed to enroll in the trial after consultation with the sponsor (Participant must also have negative urine drug screen at the screening.)
  2. A positive urine screen for drugs of abuse at screening.
  3. A history of alcohol consumption exceeding 2 standard drinks per day on average (1 glass is approximately equivalent to the following: beer [354 mL/12 oz], wine or sake [118 mL/4 oz], or distilled spirits [29.5 mL/1 oz] per day).
  4. A positive Breathalyzer test for alcohol at screening. The investigator will screen urine for drug abuse and perform an alcohol test at the inclusion visit (after consent has been signed), and may also rely on previous results obtained in the course of patient follow-up according to standard practice.
* The participant is a trial site employee, a site employee's immediate family member (for example, spouse, parent, child, sibling), or is in a dependent relationship with a site employee who is involved in conduct of this trial or may consent under duress.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 288 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2032-02-01 (Estimated); Study Completion 2032-02-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with functional remission as defined by a Personal and Social Performance Scale score >70 (minimal 1 max 100) at 24 months follow-up (study endpoint). | 24 months
  The Personal and Social Performance will be assessed at different times of the study, both by the treating psychiatrist of the patients (i.e. who is not blind to patients' treatment arm) and by the Dreams-Phen evaluation team (who will be blind to patients' treatment arm). The primary endpoint will rely ONLY on the PSP scores at 24 months assessed by the Dreams-Phen evaluation team.
  This evaluation will be performed during a webmeeting with the patient and his/her caregiver and will be based on the patient's functioning during the month preceding the evaluation.

IPD SHARING:
Plan to Share IPD: No